CLINICAL TRIAL: NCT02451631
Title: A Multi-center, Randomized, Parallel, Open Clinical Trial to Evaluate the Glycemic Control Effect of the Mobile Healthcare Service in Patients With Type 2 Diabetes Mellitus
Brief Title: The Mobile Diabetes Mgmt. Study With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Healthconnect (Industry)
Collaborators: Seoul National University Hospital (Other); Seoul National University Bundang Hospital (Other); SMG-SNU Boramae Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SB02
Record Dates: First submitted 2015-05-18; First posted 2015-05-22 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
Keywords: Mobile Application; Diabetes management
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Paper

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Traditional care (Active Comparator): Traditional care with paper(SMBG) and healthcare staff advice in office
  Interventions: Other: Traditional care with paper
- Health-On G App.+ Physician web portal (Experimental): Patient self-mgmt using Health-On G Application on smartphone; Healthcare staffs monitoring through physician web to review data
  Interventions: Device: Health-on G App. + Physician Web

INTERVENTIONS:
Other: Traditional care with paper — Healthcare staff-driven care, Diabetes mgmt. guide-book provided. Patient self-monitoring of blood glucose(SMBG) with paper.
  Arms: Traditional care
Device: Health-on G App. + Physician Web — Patients use their smart-phone or receive rental phone, and download Health-On G application. Algorithm-based personalized feedback are provided when patients' data are linked to Health-On G Application. Patient self-monitoring blood glucose data from glucometer are transferred to App. automatically by bluetooth, or input manually, check medication regimen, input food intake and exercise, and step counts are linked by Activity tracker. Personalized feedback are instantly provided based on data. Entered data are also connected to web-based physician portal. Physician web portal is provided, where they're able to review their patient's all data. Health-On G is defined as a U-Healthcare medical device consisting of gateway and decision support system.
  Arms: Health-On G App.+ Physician web portal

SUMMARY:
A Multi-center, Randomized, Parallel, Open Clinical Trial to Evaluate the Glycemic Control Effect of the Mobile Healthcare Service Using U-Healthcare Clinical Decision Support System (CDSS) and U-Healthcare Gateway in Patients with Type 2 Diabetes Mellitus

DETAILED DESCRIPTION:
The Mobile Diabetes Intervention Study is evaluating a diabetes mgmt. algorithm system by using patient mobile application and physician web-based portal. The investigators hypothesize that patient self-monitoring of blood glucose, dietary and exercise by using application and physician's remote monitoring can additional decrease of HbA1c over 6 month.

ELIGIBILITY:
Inclusion Criteria:

* 20-80 years of age
* Type 2 diabetes patients (who have taken stably oral diabetic drugs or insulin, and been doing lifestyle improvement by doctor's advice for recent over 3 months)
* in case insulin treated, patients with basal insulin once a day or premixed insulin twice a day
* HbA1c between 7.0% and 10.0%
* ability to understand and use smartphone application

Exclusion Criteria:

* type 1 diabetes or patients using insulin pump
* severe complications (stage IV,V chronic kidney failure, diabetic food complications, unstable angina pectoris, MI or stroke, surgical procedure of coronary & peripheral artery within recent 6 months)
* uncontrolled hypertension
* pregnant woman, fertile woman who will not use contraception
* unable to use application during treatment
* taking medication which can affect on glucose level
* alcohol abuse or dependency
* over 2.5 times from the upper limit of liver enzyme level
* DKA(diabetic ketoacidosis) or HHS(Hyperglycemic hyperosmolar syndrome) history during recent 6 months

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-11 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c (%) | Change from baseline to 24 weeks

SECONDARY OUTCOMES:
Change in HbA1c (%) | Change from baseline to 12 weeks
Change in SDSCA(Summary of Diabetes Self-Care Activities) | from baseline to 24 weeks
Change in WHOQOL-BREF (World Health Organization Quality Of Life-BREF) | from baseline to 24weeks
Change in FBG(Fasting Blood Glucose) | from baseline to 12weeks and 24weeks

CONTACTS AND LOCATIONS:
Overall Officials: Young Min Cho, MD.PhD, Principal Investigator — Seoul National University Hospital
Locations (3):
- South Korea (3):
  - Seoul National University Bundang Hospital, Kyunggi-do
  - Seoul National University Boramae Medical Center, Seoul
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Background] Lim S, Kang SM, Shin H, Lee HJ, Won Yoon J, Yu SH, Kim SY, Yoo SY, Jung HS, Park KS, Ryu JO, Jang HC. Improved glycemic control without hypoglycemia in elderly diabetic patients using the ubiquitous healthcare service, a new medical information system. Diabetes Care. 2011 Feb;34(2):308-13. doi: 10.2337/dc10-1447. PMID 21270188
- [Background] Kwon HS, Cho JH, Kim HS, Song BR, Ko SH, Lee JM, Kim SR, Chang SA, Kim HS, Cha BY, Lee KW, Son HY, Lee JH, Lee WC, Yoon KH. Establishment of blood glucose monitoring system using the internet. Diabetes Care. 2004 Feb;27(2):478-83. doi: 10.2337/diacare.27.2.478. PMID 14747232
- [Derived] Kim EK, Cho YM. Response to Comment on Kim et al. The Effect of a Smartphone-Based, Patient-Centered Diabetes Care System in Patients With Type 2 Diabetes: A Randomized, Controlled Trial for 24 Weeks. Diabetes Care 2019;42:3-9. Diabetes Care. 2019 Jul;42(7):e126. doi: 10.2337/dci19-0021. No abstract available. PMID 31221711
- [Derived] Kim EK, Kwak SH, Jung HS, Koo BK, Moon MK, Lim S, Jang HC, Park KS, Cho YM. The Effect of a Smartphone-Based, Patient-Centered Diabetes Care System in Patients With Type 2 Diabetes: A Randomized, Controlled Trial for 24 Weeks. Diabetes Care. 2019 Jan;42(1):3-9. doi: 10.2337/dc17-2197. Epub 2018 Oct 30. PMID 30377185